CLINICAL TRIAL: NCT02451423
Title: Phase II Study of Neoadjuvant Atezolizumab-based Immunotherapy for Patients With Urothelial Carcinoma (NEBULA)
Brief Title: Neoadjuvant Atezolizumab in Localized Bladder Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lawrence Fong (Other)
Collaborators: Genentech, Inc. (Industry); Bladder Cancer Advocacy Network (Other); Conquer Cancer Foundation (Other); National Cancer Institute (NCI) (NIH); The V Foundation (Other)
Responsible Party: Sponsor-Investigator, Lawrence Fong, Professor in Residence, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 14524; NCI-2017-01387 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP)); R01CA194511 (NIH)
Record Dates: First submitted 2015-03-04; First posted 2015-05-22 (Estimated); Results first posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Carcinoma, Transitional Cell
Keywords: Non-metastatic; Bladder
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A1: Atezolizumab (Single dose) (Experimental): Atezolizumab will be given as a neoadjuvant treatment Intravenously (IV) on Day 1 of each 21-day Cycle, for up to 1 cycle (1200mg x 1 dose)
  Interventions: Drug: Atezolizumab
- Cohort A2: Atezolizumab Monotherapy (2 doses) (Experimental): Atezolizumab will be given as a neoadjuvant treatment Intravenously (IV) on Day 1 of each 21-day Cycle, for up to 2 cycles (1200 mg x 2 doses)
  Interventions: Drug: Atezolizumab
- Cohort A3: Atezolizumab Monotherapy (3 doses) (Experimental): Atezolizumab will be given as a neoadjuvant treatment Intravenously (IV) on Day 1 of each 21-day Cycle, for up to 3 cycles (1200 mg x 3 doses)
  Interventions: Drug: Atezolizumab

INTERVENTIONS:
Drug: Atezolizumab — 1200 mg Given IV
  Other Names: MPDL3280A

SUMMARY:
This phase II trial studies the best dose of atezolizumab in treating patients with bladder cancer that has not spread to other places in the body. Immunotherapy with monoclonal antibodies may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the intratumoral immune response associated with increasing numbers of atezolizumab (MPDL3280A) treatments. (Multi-dose cohorts, Cohort A).

II. To assess the anti-tumor activity of MPDL3280A as determined by the pathologic T0 rate (pT0) at the time of cystectomy. (Expansion cohorts, Cohort A).

SECONDARY OBJECTIVES:

I. To evaluate the safety and feasibility of administering up to 3 cycles of atezolizumab pre-operatively to patients with resectable urothelial bladder cancer (Multi-dose cohorts).

II. To assess the anti--tumor activity of neoadjuvant treatment as determined by the pathologic partial response (< pT2N0) assessed at the time of radical cystectomy (Expansion cohorts).

III. To determine the 2-year relapse-free survival (RFS) rate and median RFS from time of radical cystectomy in patients treated with neoadjuvant therapy (Expansion cohorts).

IV. To determine the 2-year overall survival (OS) and median OS from time of radical cystectomy in patients treated with neoadjuvant therapy (Expansion cohorts).

V. To assess the intratumoral immune response of neoadjuvant by comparing pre-treatment transurethral resection of bladder tumor (TURBT) with post-treatment cystectomy tumor specimens (Expansion cohorts).

EXPLORATORY (CORRELATIVE) OBJECTIVES:

I. To assess for tumor-based biomarkers of response and resistance to this combination therapy using single-cell RNA sequencing (scRNA-seq) and high-dimensional flow cytometry.

II. To assess the presence of antigen-specific immune responses to a broad panel of candidate tumor antigens.

OUTLINE: This is a dose-escalation study of atezolizumab.

COHORT A: Patients receive atezolizumab intravenously (IV) over 30-60 minutes on day 1. Treatment repeats every 21 days for up to 3 doses prior to cystectomy in the absence of disease progression or unacceptable toxicity.

COHORT B: Cohort B was never opened for enrollment.

After all neoadjuvant study therapy is administered, each subject will undergo cystectomy to evaluate pathologic response to treatment and for immunologic characterization in the resected tissue. Serum and urine will be obtained as well to characterize circulating immune responses.

After completion of study treatment, patients are followed for up every 4 weeks for 12 weeks and then every 12 weeks for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1
* Histologically document transitional cell carcinoma with the presence of any of the following stages: Carcinoma in situ (CIS), high-grade Ta, any grade T1, or any grade cT2-T4, considered appropriate for radical cystectomy. Subjects with mixed histology are required to have a dominant transitional cell carcinoma (TCC) pattern.
* For subjects with non-muscle-invasive bladder cancer (NMIBC), Bacillus Calmette-Guerin (BCG) -refractory or BCG-resistant disease. BCG-refractory disease is defined as the absence of a complete response by 6 months in patients who have received induction and maintenance OR two induction courses of BCG. BCG-resistant disease is defined as persistent or recurrent disease after 2 induction courses of BCG within 1 year OR cancer recurrence within 1 year of initiation of therapy for patients who have received induction plus maintenance BCG therapy. Subjects with NMIBC must be suitable for and willing to undergo a radical cystectomy at the completion of study therapy.
* For subjects with muscle invasive disease: not suitable neoadjuvant cisplatin-based chemotherapy as determined by the following:
* Creatinine clearance less than 60ml/min. Glomerular filtration rate (GFR) should be assessed by calculation from serum/plasma creatinine (Cockcroft-Gault formula)
* Common Terminology Criteria for Adverse Events (CTCAE) Grade >/= 2 hearing loss
* CTCAE Grade >/= 2 neuropathy
* Subjects with nonmetastatic muscle-invasive bladder cancer (MIBC) not meeting the above criteria are still eligible provided the patient declines neoadjuvant cisplatin-based chemotherapy, after specific informed consent describing the known benefits of cisplatin-based chemotherapy. The reason for declining must be documented.
* Adequate bone marrow function defined as
* White Blood Cell count (WBC) > 2500 cells/mm3
* Absolute Neutrophil Count (ANC) > 1500 cells/mm3
* Hemoglobin > 9 g/dL. Patients may be transfused or receive erythropoietic treatment to meet this criterion.
* Platelet count > 100,000 cells/mm3
* Adequate renal function: Serum creatinine < 2 mg/dL OR calculated Creatinine Clearance (CrCl) > 30ml/min
* Serum bilirubin < 1.5 x ULN (except for patients with documented Gilbert's disease)
* aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2.5 x upper limit of normal (ULN)
* Ability to understand and willingness to sign a written informed consent.
* Have available evaluable archival tumor tissue for PD-L1 biomarker assessment. Presence of PD-L1 antigen on tumors is NOT required for study entry.
* The effects of MPDL3280A on the developing human fetus are unknown. For this reason women of child-bearing potential and men must agree to use adequate contraception prior to study entry, during study participation, and for 90 days after study treatment discontinuation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and for 90 days after completion of study drug administration.

Exclusion Criteria:

* Subjects with primary TCC of the ureter, urethra, or renal pelvis without TCC of the bladder are not allowed.
* Known distant metastatic disease (e.g. pulmonary or hepatic metastases).
* Subjects with malignant lymphadenectomy in the abdomen or pelvis considered appropriate for radical cystectomy and lymphadenectomy with the goal of complete resection of all malignant disease are allowed.
* Intravesical chemo- or biologic therapy within 6 weeks of first treatment.
* Prior systemic chemotherapy or radiation therapy for transitional cell carcinoma of the bladder.
* Subjects who have received prior intravesical chemotherapy are allowed.
* Prior treatment with CD137 agonists or immune checkpoint blockade therapies, including anti cytotoxic T-lymphocyte-associated protein 4 (CTLA-4), anti-programmed cell death protein 1 (PD-1) and anti-PD-L1 therapeutic antibodies.
* History of autoimmune disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegner's granulomatosis, Sjogren's syndrome, Guillain-Barre syndrome, multiple sclerosis, vacuities, or glomerulonephritis.
* Patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone are eligible for this study.
* Patients with controlled Type I diabetes mellitus on a stable dose of insulin regimen are eligible for this study.
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan.
* History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
* Chronic liver disease
* HIV or active hepatitis B virus (HBV); chronic or acute; defined as having a positive hepatitis B surface antigen [Bag] test at screening) or active hepatitis C
* Patients with past HBV infection or resolved HBV infection (defined as the presence of hepatitis B core antibody (HBcAb) and absence of HBsAg) are eligible. HBV DNA must be obtained in these patients prior to Cycle 1, Day 1, but detection of HBV DNA in these patients will not exclude study participation.
* Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Active tuberculosis
* Severe infections within 4 weeks prior to Cycle 1, Day 1, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia
* Prior allogeneic stem cell or solid organ transplant
* Administration of a live, attenuated vaccine within 4 weeks before Cycle 1, Day 1 or anticipation that such a live attenuated vaccine will be required during the study. Inactivated vaccines (such as hepatitis A or polio vaccines) are permitted during the study.
* Influenza vaccination should be given during influenza season only (approximately October to March). Patients must not receive live attenuated influenza vaccine (e.g., FluMist) within 4 weeks prior to Cycle 1, Day 1 and for at least 12 weeks after the last dose.
* Clinically significant active infection or uncontrolled medical condition
* Uncontrolled cystitis, significant bladder pain or spasms, or gross hematuria that in the opinion of the treating investigator, should preclude study entry.
* Significant cardiovascular disease, such as New York Heart Association cardiac disease (Class II or greater), myocardial infarction within the previous 3 months, unstable arrhythmias, or unstable angina
* Patients with known coronary artery disease, congestive heart failure not meeting the above criteria, or left ventricular ejection fraction < 50% must be on a stable medical regimen that is optimized in the opinion of the treating physician, in consultation with a cardiologist if appropriate.
* Major surgical procedure other than for diagnosis within 28 days prior to Cycle 1, Day 1 or anticipation of need for a major surgical procedure other than cystectomy during the course of the study
* Treatment with systemic corticosteroids or other systemic immunosuppressive medications (including but not limited to prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor (anti-TNF) agents within 2 weeks prior to Cycle 1, Day 1, or anticipated requirement for systemic immunosuppressive medications during the trial
* Patients who have received acute, low-dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea) may be enrolled in the study after discussion with and approval by the Study Chair.
* The use of inhaled corticosteroids and mineralocorticoids (e.g., fludrocortisone for adrenal insufficiency) is allowed.
* Pregnant or nursing women are excluded
* Known hypersensitivity to Chinese hamster ovary (CHO) cell products or any component of the MPDL3280A formulation
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* Malignancies other than Urological Cancers (UC) within 5 years prior to Cycle 1, Day 1, with the exception of those with a low risk of metastasis or death treated with expected curative outcome (such as, but not limited to, adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer treated with curative intent and absence of Prostate-specific antigen (PSA) relapse, or ductal carcinoma in situ of the breast treated surgically with curative intent) or incidental prostate cancer (T1a, Gleason score ≤ 6 and PSA < 0.5 ng/mL).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-03-29 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Fong, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oh DY, Kwek SS, Raju SS, Li T, McCarthy E, Chow E, Aran D, Ilano A, Pai CS, Rancan C, Allaire K, Burra A, Sun Y, Spitzer MH, Mangul S, Porten S, Meng MV, Friedlander TW, Ye CJ, Fong L. Intratumoral CD4+ T Cells Mediate Anti-tumor Cytotoxicity in Human Bladder Cancer. Cell. 2020 Jun 25;181(7):1612-1625.e13. doi: 10.1016/j.cell.2020.05.017. Epub 2020 Jun 3. PMID 32497499
- [Derived] Friebel E, Kapolou K, Unger S, Nunez NG, Utz S, Rushing EJ, Regli L, Weller M, Greter M, Tugues S, Neidert MC, Becher B. Single-Cell Mapping of Human Brain Cancer Reveals Tumor-Specific Instruction of Tissue-Invading Leukocytes. Cell. 2020 Jun 25;181(7):1626-1642.e20. doi: 10.1016/j.cell.2020.04.055. Epub 2020 May 28. PMID 32470397

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Cohort B was never opened to accrual
Groups:
- Cohort A1: Atezolizumab Monotherapy (Single Dose): Atezolizumab will be given as a neoadjuvant treatment Intravenously (IV) on Day 1 of each 21-day Cycle, for up to 1 cycle (1200mg x 1 dose)
Period: Overall Study
Arm/Group | Cohort A1: Atezolizumab Monotherapy (Single Dose) | Cohort A2: Atezolizumab Monotherapy (2 Doses) | Cohort A3: Atezolizumab Monotherapy (3 Doses)
Started | 6 | 6 | 11
Completed | 6 | 6 | 11
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A1: Atezolizumab Monotherapy (Single Dose) | Cohort A2: Atezolizumab Monotherapy (2 Doses) | Cohort A3: Atezolizumab Monotherapy (3 Doses) | Total
Number analyzed (Participants) | 6 | 6 | 11 | 23
Age, Customized [Count of Participants; unit: Participants]
  60-69 years old | 2 | 4 | 5 | 11
  70-79 years old | 3 | 2 | 6 | 11
  80-89 years old | 1 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 1 | 8
  Male | 3 | 2 | 10 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 3
  Not Hispanic or Latino | 5 | 5 | 10 | 20
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 6 | 5 | 8 | 19
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 11 | 23

OUTCOME MEASURES:

1. Primary Outcome: Mean log2 (Fold Change of CD3+ T-Cell Count/µm2) Over Time
Description: The immunologic effect MPDL3280A activity within bladder tissue will be measured by a change in the Cluster of differentiation 3 positive (CD3+) T cell count/µm2 between pretreatment biopsy and cystectomy tissue following MPDL3280A infusions. For each cohort, the mean of the log2 of ratio of post-treatment vs. pre-treatment counts with 95% confidence intervals will be reported.
Time Frame: Up to 1 year
Population: Only 12 participants had evaluable pretreatment biopsy and cystectomy tissue following MPDL3280A infusions required for this protocol endpoint.
Measure: Mean (95% Confidence Interval); unit: log2(fold change)
Arm/Group | Cohort A1: Atezolizumab Monotherapy (Single Dose) | Cohort A2: Atezolizumab Monotherapy (2 Doses) | Cohort A3: Atezolizumab Monotherapy (3 Doses)
Number analyzed (Participants) | 2 | 2 | 8
log2(fold change) | -0.036 [-3.326 to 3.253] | -0.041 [-2.184 to 2.103] | 1.516 [0.653 to 2.379]

2. Primary Outcome: Mean log2 (Fold Change of CD3+ Ki67+ Proliferative T Cell Count/µm2) Over Time
Description: The immunologic effect MPDL3280A activity within bladder tissue will be measured by a change in the CD3+ Ki67+ proliferative T cell count/µm2 between pretreatment biopsy and cystectomy tissue following MPDL3280A infusions. For each cohort, the mean of the log2 of ratio of post-treatment vs. pre-treatment counts with 95% confidence intervals will be reported.
Time Frame: Up to 1 year
Population: CD3+ Ki67+ proliferative T cell count/µm2 data was not collected.
Arm/Group | Cohort A1: Atezolizumab Monotherapy (Single Dose) | Cohort A2: Atezolizumab Monotherapy (2 Doses) | Cohort A3: Atezolizumab Monotherapy (3 Doses)
Number analyzed (Participants) | 0 | 0 | 0

3. Primary Outcome: Mean log2 (Fold Change of CD4+ FoxP3- Helper T Cell Count/µm2) Over Time
Description: The immunologic effect MPDL3280A activity within bladder tissue will be measured by a change in the cluster of differentiation 4 positive (CD4+) FoxP3- helper T cells count/µm2 between pretreatment biopsy and cystectomy tissue following MPDL3280A infusions. For each cohort, the mean of the log2 of ratio of post-treatment vs. pre-treatment counts with 95% confidence intervals will be reported.
Time Frame: Up to 1 year
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: log2(fold change)
Arm/Group | Cohort A1: Atezolizumab Monotherapy (Single Dose) | Cohort A2: Atezolizumab Monotherapy (2 Doses) | Cohort A3: Atezolizumab Monotherapy (3 Doses)
Number analyzed (Participants) | 2 | 2 | 8
log2(fold change) | 0.829 [-1.818 to 3.477] | 0.831 [-1.105 to 2.768] | 0.66 [-0.637 to 1.958]

4. Primary Outcome: Mean log2 (Fold Change of CD4+ FoxP3+ Regulatory T Cell Count/µm2) Over Time
Description: The immunologic effect MPDL3280A activity within bladder tissue will be measured by a change in the CD4+ FoxP3+ regulatory T cell count/µm2 between pretreatment biopsy and cystectomy tissue following MPDL3280A infusions. For each cohort, the mean of the log2 of ratio of post-treatment vs. pre-treatment counts with 95% confidence intervals will be reported.
Time Frame: Up to 1 year
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: log2(fold change)
Arm/Group | Cohort A1: Atezolizumab Monotherapy (Single Dose) | Cohort A2: Atezolizumab Monotherapy (2 Doses) | Cohort A3: Atezolizumab Monotherapy (3 Doses)
Number analyzed (Participants) | 2 | 2 | 8
log2(fold change) | 1.556 [0.664 to 2.447] | 2.903 [2.686 to 3.12] | 0.238 [-1.215 to 1.692]

5. Primary Outcome: Mean log2 (Fold Change of CD8+ Cytotoxic T Cell Count/µm2) Over Time
Description: The immunologic effect MPDL3280A activity within bladder tissue will be measured by a change in the cluster of differentiation 8 positive (CD8+) cytotoxic T cell count/µm2 between pretreatment biopsy and cystectomy tissue following MPDL3280A infusions. For each cohort, the mean of the log2 of ratio of post-treatment vs. pre-treatment counts with 95% confidence intervals will be reported.
Time Frame: Up to 1 year
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: log2(fold change)
Arm/Group | Cohort A1: Atezolizumab Monotherapy (Single Dose) | Cohort A2: Atezolizumab Monotherapy (2 Doses) | Cohort A3: Atezolizumab Monotherapy (3 Doses)
Number analyzed (Participants) | 2 | 2 | 8
log2(fold change) | 0.937 [-0.496 to 2.369] | 0.666 [-0.992 to 2.324] | 2.017 [0.384 to 3.65]

6. Primary Outcome: Percentage of Participants With a Treatment-related Delay
Description: The percentage of participants requiring a treatment-related delay in surgery beyond 12 weeks from study start will be summarized using descriptive statistics.
Time Frame: Up to 2 years
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A1: Atezolizumab Monotherapy (Single Dose) | Cohort A2: Atezolizumab Monotherapy (2 Doses) | Cohort A3: Atezolizumab Monotherapy (3 Doses)
Number analyzed (Participants) | 6 | 6 | 11
percentage of participants | 0 | 0 | 0

7. Primary Outcome: Number of Participants With Maximum Grade Treatment-related Toxicities Prior to Surgery
Description: Treatment-related adverse events occurring prior to surgery will be summarized by maximum toxicity grade for all participants treated with a particular regimen. The grade of toxicity will be calculated using NCI CTCAE version 4.0.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A1: Atezolizumab Monotherapy (Single Dose) | Cohort A2: Atezolizumab Monotherapy (2 Doses) | Cohort A3: Atezolizumab Monotherapy (3 Doses)
Number analyzed (Participants) | 6 | 6 | 11
Participants
  Diarrhea | 1 | 0 | 0
  Abdominal Pain | 1 | 0 | 0
  Rash maculo-papular | 0 | 1 | 2
  Musculoskeletal and connective tissue disorder - Other (Joint Ache) | 0 | 1 | 0
  Fatigue | 0 | 2 | 3
  Hematuria | 0 | 1 | 0
  Headache | 0 | 1 | 0
  Alopecia | 0 | 1 | 0
  Skin and Subcutaneous disorders, Other (Scrotal skin disruption) | 0 | 0 | 1
  Alanine aminotransferase increased | 0 | 0 | 1
  Aspartate aminotransferase increased | 0 | 0 | 1
  Chills | 0 | 0 | 1
  Creatinine increased | 0 | 0 | 2
  Weight loss | 0 | 0 | 2
  Pain | 0 | 0 | 1
  Hyponatremia | 0 | 0 | 1

8. Secondary Outcome: Near Complete Pathologic Response Rate
Description: Point estimates and 95% confidence intervals of the near complete pathologic response rate, defined as the presence of only pTa or pTis in patients with T2 or greater disease at baseline.
Time Frame: Up to 2 years
Population: One participant in Cohort A2 had T1 disease at baseline and did not meet the T2 or greater criteria for inclusion in this analysis.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Cohort A1: Atezolizumab Monotherapy (Single Dose) | Cohort A2: Atezolizumab Monotherapy (2 Doses) | Cohort A3: Atezolizumab Monotherapy (3 Doses)
Number analyzed (Participants) | 6 | 5 | 11
proportion of participants | 0.2967 [0.03005 to 0.5635] | 0 [NA to NA] — insufficient number of participants with events | 0 [NA to NA] — insufficient number of participants with events

9. Secondary Outcome: Relapse-free Survival (RFS) Rate Intention-To-Treat (ITT) Population
Description: The percentage of participants with a two- year RFS defined from study start until recurrence of disease or death from any cause, will be obtained using the Kaplan Meier method for the ITT population.
Time Frame: Up to 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A1: Atezolizumab Monotherapy (Single Dose) | Cohort A2: Atezolizumab Monotherapy (2 Doses) | Cohort A3: Atezolizumab Monotherapy (3 Doses)
Number analyzed (Participants) | 6 | 6 | 11
percentage of participants | 67 [38 to 100] | 83 [58 to 100] | 82 [62 to 100]

10. Secondary Outcome: Overall Survival Rate
Description: Overall survival rate will be reported as the percentage of participants from study start until death from any cause obtained by Kaplan Meier method for the ITT population.
Time Frame: Up to 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A1: Atezolizumab Monotherapy (Single Dose) | Cohort A2: Atezolizumab Monotherapy (2 Doses) | Cohort A3: Atezolizumab Monotherapy (3 Doses)
Number analyzed (Participants) | 6 | 6 | 11
percentage of participants | 80 [52 to 100] | 83 [59 to 100] | 100 [100 to 100]

11. Secondary Outcome: Association of Tumor and T-cell PD-L1/PD-1 Immunohistochemical Expression With Disease Response
Description: Fisher's exact test will be used to test the association of baseline tumor and T-cell programmed death-ligand 1 (PD-L1)/programmed cell death protein 1 (PD-1) immunohistochemical expression with disease response.
Time Frame: Up to 2 years
Population: Tumor and T-cell PD-L1/PD-1 immunohistochemical expression data was not collected.
Arm/Group | Cohort A1: Atezolizumab Monotherapy (Single Dose) | Cohort A2: Atezolizumab Monotherapy (2 Doses) | Cohort A3: Atezolizumab Monotherapy (3 Doses)
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | Cohort A1: Atezolizumab Monotherapy (Single Dose) | Cohort A2: Atezolizumab Monotherapy (2 Doses) | Cohort A3: Atezolizumab Monotherapy (3 Doses)
All-Cause Mortality (participants affected / at risk) | 1/6 | 1/6 | 0/11
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/6 | 0/11
Other Adverse Events (participants affected / at risk) | 6/6 | 5/6 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A1: Atezolizumab Monotherapy (Single Dose) (N=6) | Cohort A2: Atezolizumab Monotherapy (2 Doses) (N=6) | Cohort A3: Atezolizumab Monotherapy (3 Doses) (N=11)
Kidney infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Cohort A1: Atezolizumab Monotherapy (Single Dose) (N=6) | Cohort A2: Atezolizumab Monotherapy (2 Doses) (N=6) | Cohort A3: Atezolizumab Monotherapy (3 Doses) (N=11)
Fatigue (General disorders) | 2 (2) | 3/5 (3) | 3 (3)
Fever (General disorders) | 1 (1) | 0/5 (0) | 1 (1)
Localized edema (General disorders) | 1 (1) | 0/5 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1/5 (1) | 1 (1)
Chills (General disorders) | 0 (0) | 0/5 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1/5 (1) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 3 (12) | 0/5 (0) | 1 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0/5 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1/5 (1) | 0 (0)
Fecal incontinence (Gastrointestinal disorders) | 1 (1) | 0/5 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1/5 (1) | 0 (0)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 0/5 (0) | 1 (1) — Gastric hemorrhage
Malabsorption (Gastrointestinal disorders) | 1 (1) | 0/5 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (4) | 1/5 (2) | 1 (1)
Kidney infection (Infections and infestations) | 0 (0) | 0/5 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0/5 (0) | 1 (1)
Creatinine increased (Investigations) | 2 (4) | 0/5 (0) | 3 (4)
Weight loss (Investigations) | 0 (0) | 1/5 (1) | 2 (2)
Blood bilirubin increased (Investigations) | 1 (2) | 0/5 (0) | 0 (0)
Aortic injury (Injury, poisoning and procedural complications) | 0 (0) | 0/5 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0/5 (0) | 0 (0)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 (0) | 0/5 (0) | 1 (1) — Knee injury
Intestinal stoma site bleeding (Injury, poisoning and procedural complications) | 0 (0) | 0/5 (0) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 0/5 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0/5 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 2/5 (2) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1/5 (1) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0/5 (0) | 1 (1)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 (0) | 0/5 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 0/5 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0/5 (0) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0/5 (0) | 2 (4)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0/5 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (7) | 0/5 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0/5 (0) | 3 (9)
White blood cell decreased (Investigations) | 0 (0) | 0/5 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0/5 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0/5 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0/5 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0/5 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0/5 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1/5 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0/5 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 0/5 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 0/5 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 1/5 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0/5 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0/5 (0) | 0 (0)
Skin and subcutaneous tissue disorders, Other (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Scrotal skin disruption
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Joint Aches
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-29): https://cdn.clinicaltrials.gov/large-docs/23/NCT02451423/Prot_SAP_001.pdf
  • Informed Consent Form (2021-10-14): https://cdn.clinicaltrials.gov/large-docs/23/NCT02451423/ICF_000.pdf